CLINICAL TRIAL: NCT05499052
Title: Nordics and Switzerland Prospective Multicentre Non-Interventional Observational Study to Assess the Pattern of Use of REKOVELLE® in Women Undergoing In Vitro Fertilisation (IVF) or Intracytoplasmic Sperm Injection (ICSI) Procedures in Routine Clinical Practice (NORSOS)
Brief Title: Trial to Assess the Pattern of Use of REKOVELLE® in Women Undergoing In Vitro Fertilisation (IVF) or Intracytoplasmic Sperm Injection (ICSI) Procedures in Routine Clinical Practice
Acronym: NORSOS
Status: Completed | Type: Observational
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 000411
Record Dates: First submitted 2022-07-11; First posted 2022-08-12 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Controlled Ovarian Stimulation
MeSH Terms: interventions — follitropin delta

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- REKOVELLE®
  Interventions: Drug: REKOVELLE®

INTERVENTIONS:
Drug: REKOVELLE® — Subjects must be treated according to the routine clinical practice and REKOVELLE® must be prescribed in accordance with the terms of the marketing authorisation of each participating country.
  According to the label the REKOVELLE® dose should be based on a recent determination of body weight and a recent determination of Anti-Müllerian Hormone (AMH) (i.e. within the last 12 months) measured by the following diagnostic tests: ELECSYS AMH Plus immunoassay from Roche or alternatively the ACCESS AMH Advanced from Beckman Coulter or LUMIPULSE G AMH from Fujirebio.
  Other Names: follitropin delta

SUMMARY:
Study designed to observe the usage patterns, efficacy and safety of REKOVELLE® in women naive to IVF and ICSI, undergoing their first Controlled Ovarian Stimulation (COS) treatment cycle with REKOVELLE® in routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Females aged 18 years or older at enrolment
* Who have never been treated with (naïve) in vitro fertilisation (IVF) or intracytoplasmic sperm injection (ICSI) treatment using fresh or frozen ejaculated sperm from male partner or sperm donor
* Who are prescribed REKOVELLE® for the first time, using the dosing algorithm-based on AMH test result and body weight to define the 1st cycle dose regimen with REKOVELLE® according to the approved label
* Who have been informed verbally and in writing about this trial content, signed the inform consent and who do not object to their data being electronically processed

Exclusion Criteria:

* Currently participating in an interventional clinical trial in which any treatment or follow-up is mandated
* Women with a contraindication for prescription of REKOVELLE® treatment

  * Hypersensitivity to the active substance or to any of the excipients
  * Tumours of the hypothalamus or pituitary gland
  * Ovarian enlargement or ovarian cyst not due to polycystic ovarian syndrome
  * Gynaecological haemorrhages of unknown aetiology
  * Ovarian, uterine, or mammary carcinoma
  * Primary ovarian failure
  * Malformations of sexual organs incompatible with pregnancy
  * Fibroid tumours of the uterus incompatible with pregnancy
  * Pregnancy and breast feeding
* Women who undergo ovarian stimulation for fertility preservation
* Women placed under judicial protection, guardianship, or supervision
* Women who are considered as vulnerable population

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Women who are prescribed REKOVELLE® undergoing assisted reproductive technologies (ART) such as an in vitro fertilisation (IVF) or intracytoplasmic sperm injection (ICSI) cycle.
Sampling Method: Non-Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2022-08-28 (Actual); Primary Completion 2024-03-14 (Actual); Study Completion 2024-03-14 (Actual)

PRIMARY OUTCOMES:
Use of the algorithm-based individualized dosing regimen (daily dose of REKOVELLE® administered) | Up to day 1 of REKOVELLE® stimulation
  Calculated with body weight and AMH serum level to define the daily dose of REKOVELLE®
Daily dose of REKOVELLE® | From day 1 up to day 20 of REKOVELLE® stimulation
Number of days of treatment with REKOVELLE® | From day 1 up to day 20 of REKOVELLE® stimulation
REKOVELLE® Dose changes | From day 1 up to day 20 of REKOVELLE® stimulation
  Dose changes is the discretion of the investigator
Use of the Algorithm dosing Application | Up to day 1 of REKOVELLE® stimulation
  Use of the Ferring developed dosing app for the daily dose calculation by answering yes/no
Use of GnRH protocol for Lutenizing Hormone surge suppression | Up to day 10
  Defined as a choice between GnRH agonist and GnRH antagonist
Type of drug used for triggering of follicle maturation | Between Day 8 and Day 14
  Defined as a choice between hCG or GnRH
Luteal phase support | 24-72 hours after oocyte-retrieval
  Type and the length of luteal phase support is the discretion of the investigator.
  Decided as a choice between Progesterone, Oestrogen and hCG

SECONDARY OUTCOMES:
Rate of ongoing pregnancy (≥1 intrauterine viable fetus 10-11 weeks after embryo transfer) in the fresh cycle | 10-11 weeks after embryo transfer
Rate of ongoing pregnancy (≥1 intrauterine viable fetus 10-11 weeks after embryo transfer) following the fresh cycle, including also the first frozen embryo transfer | 10-11 weeks after embryo transfer
Number of oocytes retrieved | Following 1st cycle with REKOVELLE® (each cycle range is 5-20 days, average 9 days) at 34-36 hours
Number of oocytes/embryos/blastocysts frozen | Following 1st cycle with REKOVELLE® (each cycle range is 5-20 days, average 9 days) after oocyte retrieval
Number of embryos/blastocysts transferred | Following 1st cycle with REKOVELLE® (each cycle range is 5-20 days, average 9 days) after oocyte retrieval
Quality of fresh embryos or blastocysts transferred (excellent, good, fair, other) | Following 1st cycle with REKOVELLE® (each cycle range is 5-20 days, average 9 days) after oocyte retrieval
Positive signs of pregnancy (clinical pregnancy) | Following 1st cycle with REKOVELLE® (each cycle range is 5-20 days, average 9 days) Up to 5-6 weeks after embryo transfer
  Clinical pregnancy defined as least one gestational sac.
Positive signs of pregnancy (Positive Human chorionic gonadotropin (hCG) test or urine pregnancy test) | Following 1st cycle with REKOVELLE® (each cycle range is 5-20 days, average 9 days) Up to 10-11 weeks after embryo transfer
Pregnancy loss in women with embryo/blastocyst transfer (biochemical pregnancy, spontaneous/elective abortion, ectopic pregnancy, vanishing twin) | Up to 10-11 weeks after embryo transfer
  Biochemical pregnancy is defined as positive beta hCG (βhCG) test but no gestational sac is observed on later transvaginal ultrasound, or menstruation is reported.
  Spontaneous abortion is defined as positive βhCG test but all intrauterine gestational sacs without fetal heart beat as documented by ultrasound, or there are no viable fetuses observed by ultrasound.
  Elective abortion is defined as induced abortion done at the request of the woman for other than therapeutic reasons.
  Ectopic pregnancy is defined as extrauterine gestational sac with or without fetal heart beat as documented by ultrasound or surgery.
  Vanishing twin is defined as spontaneous disappearance of an intrauterine gestational sac with or without heart beat in a pregnancy where one viable fetus remains as documented by ultrasound.
Cycle cancellation before or after oocyte pick-up and reason for cycle cancellation | At consultation visit where cycle cancellation decided up to 10-11 weeks after embryo transfer
  Date when the investigator decides to cancel cycle before oocyte pick up (due to poor ovarian response, excessive ovarian response, any illness which prevents oocyte collection procedure, subject not taking hCG injection at the correct time, subject choice, other) or after oocyte pick-up (due to no oocytes collected, no oocytes fertilized, abnormal fertilization, abnormal embryo development, no embryo development, OHSS, subject choice, other)
Adverse drug reactions (ADRs) | During 1st cycle with REKOVELLE® (each cycle range is 5-20 days, average 9 days), Up to 10-11 weeks after embryo transfer.
  Adverse drug reactions (ADRs) defined by the investigator
Ovarian hyperstimulation syndrome (OHSS) (including mild/moderate/severe) | During 1st cycle with REKOVELLE® (each cycle range is 5-20 days, average 9 days), Up to 10-11 weeks after embryo transfer.
  OHSS defined by the investigator (including mild/moderate/severe)
Preventive interventions for early OHSS | During 1st cycle with REKOVELLE® (each cycle range is 5-20 days, average 9 days), Up to 10-11 weeks after embryo transfer.
  Preventive interventions decided by the investigator (Triggering of final follicular maturation with GnRH agonist and fresh embryo/blastocyst transfer or cryopreservation, Cancellation of fresh embryo/blastocyst transfer)
Assessment of overall subject experience and convenience with REKOVELLE® by the Subject Questionnaire (assessed by the subject) | 34-36 hours after final injection of 1st cycle with REKOVELLE® (average 9 days)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Compliance, Study Director — Ferring Pharmaceuticals
Locations (9):
- Denmark (5):
  - Ferring Investigational Site, Copenhagen
  - Ferring Investigational Site, Horsens
  - Ferring Investigational Site, Køge
  - Ferring Investigational Site, Odense
  - Ferring Investigational Site, Søborg
- Ferring Investigational Site, Skien, Norway
- Ferring Investigational Site, Malmo, Sweden
- Switzerland (2):
  - Ferring Investigational Site, Baden
  - Ferring Investigational Site, Basel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pinborg A, Sopa N, Ekerhovd E, Iliadis SI, Kaspersen J, Gravotta E, Quaas A. Effectiveness and safety of follitropin delta in routine clinical practice in the Nordics and Switzerland (the NORSOS study): a prospective non-interventional study. Front Endocrinol (Lausanne). 2025 Sep 5;16:1613680. doi: 10.3389/fendo.2025.1613680. eCollection 2025. PMID 40979710